CLINICAL TRIAL: NCT05549583
Title: Single Dose Crossover Comparative Bioavailability Study of Sitagliptin/Metformin 50 mg/1000 mg Film-coated Tablets in Healthy Male and Female Volunteers / Fed State
Brief Title: Comparative Bioavailability Study of Sitagliptin/Metformin 50 mg/1000 mg Tablets in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galenicum Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: GLU-P6-327
Record Dates: First submitted 2022-09-16; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Bioequivalence; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference group (Experimental): Thirty minutes after the start of the breakfast, a single dose of the Reference formulation was administered with approximately 240 mL of water at ambient temperature
  Interventions: Drug: Sitagliptin/metformin hydrochloride (HCl) 50/1000 mg film-coated tablet
- Test group (Experimental): Thirty minutes after the start of the breakfast, a single dose of the Test formulation was administered with approximately 240 mL of water at ambient temperature
  Interventions: Drug: Sitagliptin/metformin hydrochloride (HCl) 50/1000 mg film-coated tablet

INTERVENTIONS:
Drug: Sitagliptin/metformin hydrochloride (HCl) 50/1000 mg film-coated tablet — The subjects randomly received single oral dose of Sitagliptin/metformin hydrochloride (HCl) 50/1000 mg film-coated tablet

SUMMARY:
The objective of this study was to determine the bioequivalence of two different formulations of sitagliptin/ metformin after a single oral dose administration under fed conditions.

ELIGIBILITY:
The main Inclusion Criteria were:

* non- or ex-smokers
* body mass index within 18.5 kg/m2 to 30.0 kg/m2, inclusively
* no clinically significant abnormality found in the 12-lead electrocardiogram (ECG) performed at screening
* negative pregnancy test for female subjects
* healthy according to medical history, complete physical examination (including

Exclusion Criteria:

* Females who were lactating at screening
* Females who were pregnant according to the pregnancy test at screening or prior to the first study drug administration
* History of significant hypersensitivity to sitagliptin, metformin or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
* Presence of significant gastrointestinal, liver or kidney disease, or any other condition known to interfere with drug absorption, distribution, metabolism or excretion, or known to potentiate or predispose to undesired effects
* History of significant gastrointestinal, liver or kidney disease that may have affected drug bioavailability
* History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
* Presence of out-of-range cardiac interval (PR <110 msec, PR >200 msec, QRS<60 msec, QRS >110 msec and QTc >440 msec) on the ECG at screening or other clinically significant ECG abnormalities, unless deemed non-significant by the investigator
* Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (>3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
* Any clinically significant illness in the 28 days prior to the first study drug administration
* Use of any prescription drugs (with the exception of hormonal contraceptives or hormone replacement therapy) in the 28 days prior to the first study drug administration, that in the opinion of the investigator would have put into question the status of the volunteer as healthy
* Any history of tuberculosis or proven contact with tuberculosis
* Positive test result for alcohol and/or drugs of abuse at screening or prior to the first drug administration
* Positive screening results to HIV Ag/Ab Combo, Hepatitis B surface Antigen (HBsAG [B] [hepatitis B]) or Hepatitis C Virus (HCV [C]) tests
* Volunteers who had already been included in a previous group for this clinical study
* Volunteers who took sitagliptin and/or metformin in the 28 days prior to the first study drug administration
* Volunteers who took an Investigational Product in the 28 days prior to the first study drug administration
* Volunteers who donated 50 mL or more of blood in the 28 days prior to the first study drug administration
* Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the 56 days prior to the first study drug administration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 48 hours
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC) 0-t | 48 hours
  Evaluation of plasma concentration-time curve from zero to the time of the last measurable time point t

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs), abnormal clinical laboratory test results, physical examination findings and glycemia. | 1 week
  Adverse events were classified by System Organ Class (SOC) and Preferred Term (PT) using the Medical Dictionary for Regulatory Activities (MedDRA), version 20.1 (Medrio database) and graded as mild, moderate, or severe.
  The principal investigator or qualified designee determined the relationship of any AE to the investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma, Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schnaars Y, Gaikwad S, Gottwald-Hostalek U, Uhl W, Ribot O, Varanasi KVS, Rodriguez L, Torrejon J, Gomez L. Bioequivalence Evaluation in Healthy Volunteers: New Generic Formulations of Sitagliptin and Sitagliptin-Metformin Fixed-Dose Combination Compared with the Originator Products. Diabetes Ther. 2023 Feb;14(2):347-362. doi: 10.1007/s13300-022-01349-2. Epub 2022 Dec 16. PMID 36526947